CLINICAL TRIAL: NCT03575104
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Polysomnography Study to Assess the Efficacy and Safety of ACT-541468 in Adult and Elderly Subjects With Insomnia Disorder
Brief Title: Study to Assess the Efficacy and Safety of ACT-541468 (Daridorexant) in Adult and Elderly Subjects Suffering From Difficulties to Sleep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-078A302
Record Dates: First submitted 2018-05-17; First posted 2018-07-02 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Daridorexant 10 mg (Experimental)
  Interventions: Drug: Daridorexant
- Daridorexant 25 mg (Experimental)
  Interventions: Drug: Daridorexant
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Daridorexant — Daridorexant will be administered as tablets, orally, once daily in the evening.
  Arms: Daridorexant 10 mg; Daridorexant 25 mg
Other: Placebo — Matching placebo will be administered as tablets, orally, once daily in the evening.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess efficacy and safety of ACT-541468 (daridorexant) in adult and elderly subjects with insomnia disorder. Efficacy will be evaluated on objective and subjective sleep parameters.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure;
* Male or female aged ≥ 18 years;
* Insomnia disorder according to DSM-5 criteria;
* Insomnia Severity Index score ≥ 15;
* Insufficient sleep quantity as collected subjectively in the sleep diary and validated objectively by polysomnography;
* Women of childbearing potential must have a negative and urine pregnancy test and use the contraception scheme up to at least 30 days after last study treatment intake.

Exclusion Criteria:

* Body mass index below 18.5 or above 40.0 kg/m2;
* Any lifetime history of of related breathing disorder, periodic limb movement disorder, restless legs syndrome, circadian rhythm disorder, rapid eye movement (REM) behavior disorder, narcolepsy, or apnea/hypopnea;
* Cognitive behavioral therapy (CBT) only allowed if, the treatment started at least 1 month prior to Visit 3 and the subject agrees to continue this CBT throughout the study;
* Self-reported usual daytime napping ≥ 1 hour per day and ≥ 3 days per week;
* Acute or unstable psychiatric conditions diagnosed by the Mini International Neuropsychiatric Interview;
* Mini Mental State Examination (MMSE) score < 25 in subjects ≥ 50 years;
* For female subjects: pregnant, lactating or planning to become pregnant during projected duration of the study;
* History or clinical evidence of any disease or medical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the study assessments.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 924 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (86):
- United States (37):
  - Pulmonary Associates, Pa, Glendale, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Core Healthcare Group, Cerritos, California
  - Artemis Institute For Clinical Research - Riverside, Riverside, California
  - Pacific Research Network, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Empire Clinical Research, Upland, California
  - Innovative Clinical Research, Lafayette, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Clinical Trials Research, Lincoln, Florida
  - Clinical Research Group of St. Petersburgh, St. Petersburg, Florida
  - Neurotrials Research Incorporated, Atlanta, Georgia
  - Sleep Practitioners, LLC, Macon, Georgia
  - Hawaii Pacific Neurosciences, Honolulu, Hawaii
  - Saltzer Clinical Research, Nampa, Idaho
  - Rowe Neurology Institute, Lenexa, Kansas
  - Sleep Disorders Center of the Mid-Atlantic, Glen Burnie, Maryland
  - Neurocare Inc., Newton, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Garden City Asthma and Sleep Center, Garden City, New York
  - Research Carolina of Hickory, Hickory, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Clinical Trials of America - NC, LLC, Winston-Salem, North Carolina
  - CTI Clinical Research II, Cincinnati, Ohio
  - Ohio Sleep Medicine Institue, Dublin, Ohio
  - Cleveland Sleep Research Center, Middleburg Heights, Ohio
  - Robert V. Sibilia, MD, Inc., Wooster, Ohio
  - Brian Abaluck LLC, Paoli, Pennsylvania
  - Wesley Neurology Clinic Pc (Multiple Sclerosis), Cordova, Tennessee
  - FutureSearch Trials of Neurology, LP, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Jacksonville Center for Clinical Research, Jacksonville, Texas
  - Dm Clinical Research / Martin Diagnostic Clinic, Tomball, Texas
- Belgium (4):
  - HOSPITAL AZ SINT-JAN_Neurology department, Bruges
  - Hospital Universitair Zieknhuis Brussel, Pneumology and Sleep Laboratory, Brussels
  - University Hospital Gent, Department of General Internal Medicine and Center of neurophysiological Monitoring, Ghent
  - Hospital UZ Leuven_ Pneumology Department, Leuven
- Acibadem City Clinic Tokuda Hospital EAD, Sofia, Bulgaria
- Canada (6):
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Queensway Sleep Lab Sleep Clinic (MedSleep)- 5359 Dundas Street West, Suite 202, Etobicoke, ON M9B 1B1, Etobicoke
  - The Medical Arts Health Research Group, Kelowna
  - Somni Research Inc., Markham
  - Somni Research, Calgary, Toronto
  - CANADIAN PHASE ONWARD INC. (Toronto), Toronto
- Czechia (3):
  - Nemocnice České Budějovice, Centrum pro poruchy spánku a spánkovou medicínu, České Budějovice
  - Narodni Ustav Dusevniho Zdravi (National Institute of Mental Health), Klecany
  - Fakultní nemocnice Ostrava, Spánková laboratoř, Ostrava-Poruba
- Finland (4):
  - Vitalmed Uniklinikka, Helsinki
  - Oivauni Oy - Kuopio, Kuopio
  - Oivauni Oy - Tampere, Tampere
  - Unitutkimusyksikkö, Turun Yliopisto, Turku
- France (3):
  - CHRU De Lille - Hospital Salengro - Neurophysiologie Clinique, Lille
  - Clinique beau soleil - Department Sleep and Neurology, Montpellier
  - CHU NIMES - Unité de Sommeil, Nîmes
- Germany (12):
  - Advanced Sleep Research GmbH, Berlin
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Charité - Universitätsmedizin Berlin - Campus Benjamin Franklin Kompetenzzentrum Schlafmedizin, Berlin
  - Synexus Clinical Research GmbH, Bochum
  - Klinische Forschung Dresden GmbH, Dresden
  - Synexus Clinical Research GmbH, Frankfurt
  - Klinische Forschung Hannover Mitte GmbH, Hanover
  - Interdisziplinäre Schlafmedizin, Pfalzklinikum, Klingenmünster
  - Zentrum für Integrative Psychiatrie (ZiP) Universität zu Lübeck, Lübeck
  - Central Insitute of Mental Health Sleep laboratory Medical Faculty Mannheim/Heidelberg University, Mannheim
  - Klinik und Poliklinik für Psychiatrie, Psychosomatik und Psychotherapie der Universität am Bezirksklinikum Regensburg, Regensburg
  - SOMNIBENE Institut für Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin
- Hungary (2):
  - Magyar Honvédség Egészségügyi Központ, Neurológiai Osztály, Budapest
  - Somnius Kft. SomnoCenter Szeged, Szeged
- South Korea (10):
  - Dong-A University Hospital, Busan
  - 4F Neuroimaging analysis laboratory, 56 Dalseong-ro, Jung-gu, Daegu
  - Chungnam National University Hospital, Daejeon
  - 3F, 2nd Building, Psychiatry Outpatient, Family Counseling Room, 42 Jebong-ro, Donggu, Gwangju
  - 8F Sleep Lab, 1st Building,82, Gumi-ro 173 Beon-gil, Bundang-gu, Seongnam
  - 3F Sleep Medicine Center, 101 Daehak-Ro Jongno-Gu, Seoul
  - 1st CRC room, 2F, Jejoong building, 50-1 Yonsei-ro,, Seodaemun-gu, Seoul
  - B2F, Clinical Trial Center, Konkuk University Medical Center 120-1, Neungdong-ro, Gwangjin-gu, Seoul
  - B1F Neurological examination room, 892 Dongnam-ro, Gangdong-gu, Seoul
  - 2F Psychiatry Outpatient, 93, Jungbu-daero, Paldal-gu, Suwon
- Sweden (4):
  - Göteborgs Universitet, Centrum för sömn och vakenhetsstörningar, Gothenburg
  - Universitetssjukhuset Örebro Neurokliniken, Sömnenheten, Örebro
  - SOPHIAHEMMET (Stockholm), Stockholm
  - Sömnutredningsmottagningen, smärtcentrum Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hudgens S, Phillips-Beyer A, Newton L, Seboek Kinter D, Benes H. Development and Validation of the Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ). Patient. 2021 Mar;14(2):249-268. doi: 10.1007/s40271-020-00474-z. Epub 2020 Nov 1. PMID 33131027
- [Result] Mignot E, Mayleben D, Fietze I, Leger D, Zammit G, Bassetti CLA, Pain S, Kinter DS, Roth T; investigators. Safety and efficacy of daridorexant in patients with insomnia disorder: results from two multicentre, randomised, double-blind, placebo-controlled, phase 3 trials. Lancet Neurol. 2022 Feb;21(2):125-139. doi: 10.1016/S1474-4422(21)00436-1. PMID 35065036
- [Derived] Di Marco T, Djonlagic I, Dauvilliers Y, Sadeghi K, Little D, Datta AN, Hubbard J, Hajak G, Krystal A, Olivieri A, Parrino L, Puryear CB, Zammit G, Donoghue J, Scammell TE. Effect of daridorexant on sleep architecture in patients with chronic insomnia disorder: a pooled post hoc analysis of two randomized phase 3 clinical studies. Sleep. 2024 Nov 8;47(11):zsae098. doi: 10.1093/sleep/zsae098. PMID 38644625
- [Derived] Citrome L, Juday TR, Lundwall C. Lemborexant and Daridorexant for the Treatment of Insomnia: An Indirect Comparison Using Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. J Clin Psychiatry. 2023 Oct 2;84(6):23m14851. doi: 10.4088/JCP.23m14851. PMID 37796657
- [Derived] Dutta S, Singhal S, Shah R, Charan J, Dhingra S, Haque M. Daridorexant as a novel pharmacotherapeutic approach in insomnia: a systematic review and meta-analysis. Expert Opin Drug Saf. 2023 Jul-Dec;22(12):1237-1251. doi: 10.1080/14740338.2023.2243217. Epub 2023 Aug 7. PMID 37526060
- [Derived] Heidenreich S, Ross M, Chua GN, Seboek Kinter D, Phillips-Beyer A. Preferences of patients for benefits and risks of insomnia medications using data elicited during two phase III clinical trials. Sleep. 2022 Nov 9;45(11):zsac204. doi: 10.1093/sleep/zsac204. PMID 36054921

RESULTS

PARTICIPANT FLOW:
Groups:
- Daridorexant 10 mg; Daridorexant 25 mg: Daridorexant was administered as tablets, orally, once daily in the evening.
- Placebo: Matching placebo was administered as tablets, orally, once daily in the evening.
Period: Overall Study
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Started | 307 | 309 | 308
Completed | 283 | 280 | 286
Not Completed | 24 | 29 | 22
Not completed — Adverse Event | 4 | 3 | 4
Not completed — Withdrawal by Subject | 13 | 16 | 11
Not completed — Other reasons | 6 | 8 | 6
Not completed — Lost to Follow-up | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo | Total
Number analyzed (Participants) | 307 | 309 | 308 | 924
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 186 | 188 | 187 | 561
  >=65 years | 121 | 121 | 121 | 363
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (14.0) | 56.3 (14.4) | 56.7 (14.1) | 56.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 218 | 205 | 638
  Male | 92 | 91 | 103 | 286
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 16 | 47
  Not Hispanic or Latino | 288 | 295 | 290 | 873
  Unknown | 1 | 0 | 1 | 2
  Not permitted as per legislation/regulation | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 16 | 26 | 29 | 71
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1 | 2
  Asian | 14 | 11 | 10 | 35
  White | 273 | 271 | 267 | 811
  Not permitted as per legislation/regulation | 1 | 0 | 1 | 2
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 1 in Wake After Sleep Onset (WASO) (Sleep Maintenance)
Description: "Wake After Sleep Onset" is the time spent awake after onset of persistent sleep until lights on, as determined by polysomnography.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
minutes | -15.31 [-19.531 to -11.087] | -24.19 [-28.466 to -19.911] | -12.57 [-16.817 to -8.323]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in WASO (min) to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other — The Type I error rate was controlled for the testing of multiple null hypotheses associated with the endpoint assessed at 1 and 3 months of treatment and the two dose levels studied. Each null hypothesis was tested against the alternative hypothesis that daridorexant improved the endpoint at the given dose and time point compared to placebo. The order of testing and the alpha level applied to each null hypothesis was based on the Bonferroni-based gatekeeping procedure (see SAP for details); p = 0.0001, Mixed Models Analysis — Mixed effects model for repeated measures: change from baseline in WASO = baseline WASO + age group (< 65; ≥ 65 years) + treatment + visit + treatment × visit + baseline × visit; Hypothesis testing result: threshold for significance p = 0.025; statistically significant = YES; LS mean difference to placebo = -11.62, 95% CI 2-sided [-17.604 to -5.633]
Statistical Analysis 2: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in WASO (min) to Month 1 (Daridorexant 10 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3669, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Hypothesis testing result: threshold for significance p = 0.00977; statistically significant = NO; LS mean difference to placebo = -2.74, 95% CI 2-sided [-8.693 to 3.215]

2. Primary Outcome: Change From Baseline to Month 3 in Wake After Sleep Onset (WASO)
Description: as for outcome 1
Time Frame: From baseline to Month 3 (i.e. for up to 3 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
minutes | -15.95 [-20.734 to -11.165] | -24.25 [-29.021 to -19.474] | -14.00 [-18.756 to -9.241]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in WASO (min) to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0028, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Hypothesis testing result: threshold for significance p = 0.01563; statistically significant = YES; LS Mean difference to placebo = -10.25, 95% CI 2-sided [-16.95 to -3.548]
Statistical Analysis 2: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in WASO (min) to Month 3 (Daridorexant 10 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5686, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Hypothesis testing result: threshold for significance p = 0; statistically significant = NO; LS Mean difference to placebo = -1.95, 95% CI 2-sided [-8.666 to 4.764]

3. Primary Outcome: Change From Baseline to Month 1 in Latency to Persistent Sleep (LPS) (Sleep Onset)
Description: "Latency to Persistent Sleep" is the time from start of recording to the beginning of the first continuous 20 epochs (i.e., 10 minutes) scored as non-awake, i.e., epochs scored as either sleep stage 1 (S1), sleep stage 2 (S2), sleep stage 3 (slow wave sleep) or REM, as determined by polysomnography.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
minutes | -22.62 [-26.733 to -18.503] | -26.46 [-30.626 to -22.292] | -20.01 [-24.148 to -15.875]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in LPS (min) to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0303, Mixed Models Analysis — Mixed effects model for repeated measures: change from baseline in LPS = baseline LPS + age group (< 65; ≥ 65 years) + treatment + visit + treatment × visit + baseline × visit; Hypothesis testing result: threshold for significance p = 0.025; statistically significant = NO; LS mean difference to placebo = -6.45, 95% CI 2-sided [-12.282 to -0.614]
Statistical Analysis 2: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in LPS (min) to Month 1 (Daridorexant 10 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3782, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Hypothesis testing result: threshold for significance p = 0.00195; statistically significant = NO; LS mean difference to placebo = -2.61, 95% CI 2-sided [-8.41 to 3.197]

4. Primary Outcome: Change From Baseline to Month 3 in Latency to Persistent Sleep (LPS)
Description: as for outcome 3
Time Frame: From baseline to Month 3 (i.e. for up to 3 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
minutes | -23.09 [-27.600 to -18.571] | -28.91 [-33.413 to -24.399] | -19.89 [-24.384 to -15.405]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in LPS (min) to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0053, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Hypothesis testing result: threshold for significance p = 0.00313; statistically significant = NO; LS mean difference to placebo = -9.01, 95% CI 2-sided [-15.339 to -2.684]
Statistical Analysis 2: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in LPS (min) to Month 3 (Daridorexant 10 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3233, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Hypothesis testing result: threshold for significance p = 0; statistically significant = NO; LS mean difference to placebo = -3.19, 95% CI 2-sided [-9.528 to 3.146]

5. Secondary Outcome: Change From Baseline to Month 1 in the Subjective Total Sleep Time (sTST)
Description: "Subjective Total Sleep Time" is the total sleep time reported by the participant in the sleep diary questionnaire. A positive change from baseline indicates an increase in the subjective Total Sleep Time. A negative change from baseline indicates a decrease in subjective Total Sleep Time.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
minutes | 41.01 [35.439 to 46.584] | 43.77 [38.136 to 49.412] | 27.64 [22.015 to 33.274]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in sTST (min) to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p < .0001, Mixed Models Analysis — Hypothesis testing result: threshold for significance p = 0.0125; statistically significant = YES; LS mean difference to placebo = 16.13, 95% CI 2-sided [8.224 to 24.035]
Statistical Analysis 2: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in sTST (min) to Month 1 (Daridorexant 10 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0009, Mixed Models Analysis — Mixed effects model for repeated measures: change from baseline in sTST = baseline sTST + age group (< 65; ≥ 65 years) + treatment + visit + treatment × visit + baseline × visit; Hypothesis testing result: threshold for significance p = 0; statistically significant = NO; LS mean difference to placebo = 13.37, 95% CI 2-sided [5.507 to 21.226]

6. Secondary Outcome: Change From Baseline to Month 3 in the Subjective Total Sleep Time (sTST)
Description: Subjective Total Sleep Time is the total sleep time reported by the participant in the sleep diary questionnaire. A positive change from baseline indicates an increase in the subjective Total Sleep Time. A negative change from baseline indicates a decrease in subjective Total Sleep Time.
Time Frame: From baseline to Month 3 (i.e. for up to 3 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
minutes | 50.70 [44.398 to 57.008] | 56.18 [49.812 to 62.547] | 37.12 [30.776 to 43.464]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in sTST (min) to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; Hypothesis testing result: threshold for significance p = 0.00781; statistically significant = YES; LS mean difference to placebo = 19.06, 95% CI 2-sided [10.125 to 27.994]
Statistical Analysis 2: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in sTST (min) to Month 3 (Daridorexant 10 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0028, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; Hypothesis testing result: threshold for significance p = 0; statistically significant = NO; LS mean difference to placebo = 13.58, 95% CI 2-sided [4.691 to 22.475]

7. Secondary Outcome: Change From Baseline to Month 1 in Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ) Sleepiness Domain Score
Description: The Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ) is a validated patient reported outcome instrument comprising 14 items (each using a numeric rating scale from 0 to 10) grouped into three domains (i.e., sleepiness, mood, and alert/cognition) reflecting daytime impairment of insomnia. The IDSIQ sleepiness domain has 4 items, and the domain score ranges from 0 to a maximum of 40, where a higher score indicates a greater burden. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
Scores on a scale | -3.18 [-3.763 to -2.599] | -3.51 [-4.096 to -2.917] | -2.75 [-3.340 to -2.163]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in IDSIQ sleepiness domain score to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0733, Mixed Models Analysis — Mixed effects model for repeated measures: change from baseline in IDSIQ sleepiness domain score = baseline IDSIQ sleepiness domain score + age group (< 65; ≥ 65 years) + treatment + visit + treatment × visit + baseline × visit; Hypothesis testing result: threshold for significance p = 0.00625; statistically significant = NO; LS mean difference to placebo = -0.75, 95% CI 2-sided [-1.581 to 0.071]
Statistical Analysis 2: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in IDSIQ sleepiness domain score to Month 1 (Daridorexant 10 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3048, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Hypothesis testing result: threshold for significance p = 0; statistically significant = NO; LS mean difference to placebo = -0.43, 95% CI 2-sided [-1.251 to 0.392]

8. Secondary Outcome: Change From Baseline to Month 3 in IDSIQ Sleepiness Domain Score
Description: as for outcome 7
Time Frame: From baseline to Month 3 (i.e. for up to 3 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
Scores on a scale | -4.75 [-5.437 to -4.056] | -5.27 [-5.964 to -4.569] | -4.01 [-4.705 to -3.322]
Statistical Analysis 1: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in IDSIQ sleepiness domain score to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0120, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Hypothesis testing result: threshold for significance p = 0.00391; statistically significant = NO; LS mean difference to placebo = -1.25, 95% CI 2-sided [-2.230 to -0.276]
Statistical Analysis 2: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in IDSIQ sleepiness domain score to Month 3 (Daridorexant 10 mg vs placebo); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1393, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Hypothesis testing result: threshold for significance p = 0; statistically significant = NO; LS mean difference to placebo = -0.73, 95% CI 2-sided [-1.706 to 0.239]

9. Post Hoc Outcome: Change From Baseline to Month 1 in Log-transformed LPS (LSGM Ratio to Baseline)
Description: Post-hoc analyses were performed using log-transformed LPS data, as the LPS values at baseline more closely resembled a log-normal distribution (skewed to the right) than a normal distribution.
Time Frame: From baseline to Month 1 (i.e. for up to 1 month)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
minutes | 0.59 [0.54 to 0.64] | 0.50 [0.46 to 0.55] | 0.63 [0.58 to 0.69]
Statistical Analysis 1: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in log transformed LPS (min) to Month 1 (Daridorexant 10 mg vs placebo); Test type: Other; p = 0.2506, Mixed Models Analysis — Mixed effects model for repeated measures: log(value/baseline) = log(baseline) + age group(< 65; ≥ 65 years) + treatment + visit + treatment x visit + log(baseline) x visit; LS mean difference to placebo = 0.93, 95% CI 2-sided [0.82 to 1.05]
Statistical Analysis 2: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in log transformed LPS (min) to Month 1 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0004, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; LS mean difference to placebo = 0.80, 95% CI 2-sided [0.71 to 0.91]

10. Post Hoc Outcome: Change From Baseline to Month 3 in Log-transformed LPS (LSGM Ratio to Baseline)
Description: as for outcome 9
Time Frame: From baseline to Month 3 (i.e. for up to 3 month)
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 308
minutes | 0.56 [0.51 to 0.61] | 0.48 [0.43 to 0.52] | 0.58 [0.53 to 0.64]
Statistical Analysis 1: Comparison: Daridorexant 10 mg vs Placebo; Between-treatment analysis for change from baseline in log transformed LPS (min) to Month 3 (Daridorexant 10 mg vs placebo); Test type: Other; p = 0.5037, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; LS mean difference to placebo = 0.96, 95% CI 2-sided [0.84 to 1.09]
Statistical Analysis 2: Comparison: Daridorexant 25 mg vs Placebo; Between-treatment analysis for change from baseline in LPS (min) to Month 3 (Daridorexant 25 mg vs placebo); Test type: Other; p = 0.0021, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; LS mean difference to placebo = 0.81, 95% CI 2-sided [0.71 to 0.93]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were AEs that started or worsened on or after the DB study treatment start date up to the earlier of 30 days after DB study treatment end date or the date of enrollment in the ID-078A303 extension study. The planned duration of DB treatment was 84 days ± 2 days, i.e., 12 weeks ± 2 days.
Description: The number of subjects affected is the number of subjects with at least one event.
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/306 | 0/308 | 0/306
Serious Adverse Events (participants affected / at risk) | 3/306 | 3/308 | 4/306
Other Adverse Events (participants affected / at risk) | 49/306 | 28/308 | 30/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daridorexant 10 mg (N=306) | Daridorexant 25 mg (N=308) | Placebo (N=306)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daridorexant 10 mg (N=306) | Daridorexant 25 mg (N=308) | Placebo (N=306)
Headache (Nervous system disorders) | 14 (19) | 16 (16) | 11 (12)
Nasopharyngitis (Infections and infestations) | 38 (41) | 13 (15) | 20 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Idorsia for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, Idorsia may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (2):
  • Study Protocol (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT03575104/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03575104/SAP_001.pdf